CLINICAL TRIAL: NCT05155839
Title: An Open-label, Multicenter, First-in-human, Phase I Dose-escalation and Expansion Clinical Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of MRG001 in Patients With CD20-positive Relapsed or Refractory B-cell Non-Hodgkin Lymphoma (NHL)
Brief Title: Safety and Preliminary Efficacy Study of MRG001 in Patients With Non-Hodgkin Lymphoma (NHL)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Miracogen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRG001-001
Record Dates: First submitted 2021-12-01; First posted 2021-12-14 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Relapsed or Refractory B-cell Non-Hodgkin Lymphoma (NHL)
Keywords: MRG001; Antibody Drug Conjugate (ADC); CD20; Non-Hodgkin lymphoma (NHL)
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRG001 (Experimental): All patients in Phase Ia (dose escalation) and Phase Ib (dose expansion) will be administrated MRG001 on Day 1 of every 3 weeks (21-day cycle).
  Interventions: Drug: MRG001

INTERVENTIONS:
Drug: MRG001 — Administrated intravenously

SUMMARY:
This study consists of two parts. Phase Ia is a dose escalation study to determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of MRG001. Phase Ib is a dose expansion study to assess the preliminary efficacy of MRG001 in patients with CD20-positive relapsed or refractory B-cell NHL at the confirmed RP2D. The safety, tolerability, pharmacokinetic (PK) and immunogenicity of MRG001 will be evaluated in both parts.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participates in the clinical study; Fully understands and informed of this study, and provides written informed consent; Willing to follow and have the ability to complete all trial procedures.
2. Aged 18 to 80 (including 18 and 80), male or female.
3. Patients with histopathologically confirmed relapsed/refractory B-cell non-Hodgkin lymphoma.
4. Relapsed or refractory disease after standard of care treatment with anti-CD20 antibodies.
5. Patients must have at least one measurable lesion without prior local therapy according to Lugano 2014 criteria.
6. The score of ECOG for performance status is 0 or 1.
7. Patients without severe hematopoietic, liver and kidney dysfunction.
8. Expected survival time ≥ 3 months.
9. Prior anti-tumor treatment-related AEs (NCI CTCAE v5.0 Criteria) have recovered to ≤ Grade 1.
10. Negative blood pregnancy test for women of childbearing potential within 7 days prior to the first dose of study drug. Patients of childbearing potential should agree to use effective contraception from signing the ICF until 3 months after the last dose of study drug.
11. The score of left ventricular ejection fraction (LVEF) is > 50%.

Exclusion Criteria:

1. Applicable to Phase Ia: positive hepatitis B surface antigen (HBsAg), or negative HBsAg with a peripheral blood hepatitis B virus DNA copy number greater than the upper limit of normal; positive hepatitis C virus (HCV) antibody and positive HCV RNA at screening. Patients with a history of clinically significant non-viral hepatitis and cirrhosis. Applicable to Phase Ib: positive hepatitis B surface antigen (HBsAg) and/or positive hepatitis B core antibody (HBcAb) at screening, and peripheral blood hepatitis B virus DNA copy number greater than the upper limit of normal; positive hepatitis C virus (HCV) antibody and positive HCV RNA. Patients with a history of clinically significant non-viral hepatitis and cirrhosis (decompensated cirrhosis Child-Pugh class B, C).
2. Positive human immunodeficiency virus (HIV) antibody.
3. Any active infection requiring systemic therapy occurred within 2 weeks before enrollment.
4. Suspected or confirmed central nervous system invasion of NHL.
5. Allergic constitution or known hypersensitivity to rituximab or other anti-CD20 monoclonal antibodies and their components, or hypersensitivity to any component of MRG001.
6. Patients with uncontrolled or significant cardiovascular disease.
7. History of severe pulmonary disease.
8. Received CAR-T therapy within 3 months before enrollment.
9. Received blood transfusion within 28days before enrollment, or receiced erythropoietin (EPO), granulocyte colony-stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF) and other drugs that may affect hemogram within 14 days before enrollment.
10. Current use of potent CYP3A4 inhibitors or inducers.
11. History of allogeneic stem cell transplantation or organ transplantation, or have received autologous stem cell transplantation within 3 months prior to screening, or plan to undergo stem cell transplantation.
12. Suffered from other malignancies within the last 5 years.
13. Major surgery within 6 weeks prior to enrollment or planned major surgery within the first 12 weeks after receiving study drug.
14. Patients who are receiving any approved or investigational anti-tumor treatment with antibody/fusion protein/ADC drugs, radiotherapy, chemotherapy, Chinese patent medicine or Chinese herbal medicine within 28 days before enrollment; or have participated in any approved or investigational small molecule targeted therapy within 28 days before enrollment or within 5 half-lives (whichever is shorter).
15. Received any vaccine within 28 days prior to enrollment or will receive any vaccine within 6 months after the last dose of study drug.
16. Requires treatment with glucocorticoids or other immunosuppressive agents for a certain condition within 14 days prior to enrollment.
17. An acute oncolytic reaction may occur at the discretion of the investigator.
18. Inability to complete protocol-specified study visits and study drug administration.
19. Women during pregnancy or lactation; men and women of childbearing potential who are unwilling to take prescribed appropriate contraceptive measures.
20. Other conditions inappropriate for participation in this clinical trial at the discretion of the investigator.
21. Malignant lymphoma with pathological transformation.
22. High-grade B-cell lymphoma.
23. Patient's Body Mass Index ≤ 17 kg/m2.
24. Patients with underlying medical conditions that, in the judgment of the investigator, might increase the risk of receiving study drug or might affect the safety assessment of the study drug.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2019-06-25 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Baseline to 90 days after the last dose of study treatment.
  Any reaction, side effect, or untoward event that occurs during the course of the clinical trial whether or not the event is considered related to the study drug.
Maximum Tolerated Dose (MTD) | DLT will be evaluated during the first treatment cycle (Day 1-21).
  The highest dose confirmed wherein ≤ 1/6 of patients in a treatment cohort experiences a dose-limiting toxicity (DLT) within 21 days after the first dose of study treatment.
Recommended Phase II Dose (RP2D) | Baseline to study completion (up to 15 months).
  The dose level of MRG001 recommended for further phase II clinical studies.

SECONDARY OUTCOMES:
PK parameter: Concentration-time curve | Baseline to 90 days after the last dose of study treatment.
  Plot of drug concentration changing with time after drug administration.
Immunogenicity | Baseline to 30 days after the last dose of study treatment
  The proportion of patients with positive ADA immunogenicity results.
Objective Response Rate (ORR) | Baseline to study completion (up to 15 months)
  ORR is defined as the proportion of subjects with CR and PR.
Duration of Response (DoR) | Baseline to study completion (up to 15 months)
  DoR is defined as the duration from the initial recording of objective disease response to the first onset of tumor progression, or death of any cause.
Disease Control Rate (DCR) | Baseline to study completion (up to 15 months)
  DCR is defined as the percentage of patients who achieve CR, PR, and stable disease (SD) after treatment.
Progression Free Survival (PFS) | Baseline to study completion (up to 15 months)
  PFS is defined as the duration from the start of treatment to the onset of tumor progression or death of any cause.
Overall Survival (OS) | Baseline to study completion (up to 15 months)
  OS is defined as the duration from the start of treatment to death of any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, Doctor, Principal Investigator — Peking University Cancer Hospital & Institute; Yuqing Song, Doctor, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (12):
- China (12):
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Hospital, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Harbin First Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No